CLINICAL TRIAL: NCT05041673
Title: Efficacy of Vildagliptin, Liraglutide and Empagliflozin in the Management of Fatty Liver Disease Among Patients With Type 2 Diabetes
Brief Title: Anti-diabetic Drugs and Fatty Liver Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Collaborators: Eva Pharma (Industry)
Responsible Party: Principal Investigator, Ahmed Kamal, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0304932
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Fatty Liver, Nonalcoholic; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Metformin; Liraglutide; empagliflozin; Vildagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): metformin +/- insulin +/- sulfonylurea
  Interventions: Drug: Metformin
- Group 2 (Experimental): Metformin plus vildagliptin +/- insulin +/- sulfonylurea
  Interventions: Drug: Metformin
- Group 3 (Experimental): Metformin plus liraglutide +/- insulin+/- sulfonylurea
  Interventions: Drug: Metformin
- Group 4 (Experimental): Metformin plus empagliflozin +/- insulin +/- sulfonylurea
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Antidiabetic drugs
  Other Names: Liraglutide; empagliflozin; Vildagliptin

SUMMARY:
Type 2 DM is one of the major risk factors for development of non-alcoholic fatty liver disease. The pooled prevalence of fatty liver among diabetics is 54% (95% CI 45%-64%). Until now there is no well-established treatment for fatty liver disease.

Study setting: Randomized controlled trial

Study population:

Patients with type 2 DM plus Fatty Liver.

Arms and Interventions

1. Experimental arms: Group 1: metformin +/- insulin +/- sulfonylurea Group 2: Metformin plus vildagliptin+/- insulin +/- sulfonylurea Group 3: Metformin plus liraglutide+/- insulin+/- sulfonylurea Group 4: Metformin plus empagliflozin +/- insulin +/- sulfonylurea

DETAILED DESCRIPTION:
Rational: Type 2 DM is one of the major risk factors for development of non-alcoholic fatty liver disease. The pooled prevalence of fatty liver among diabetics is 54% (95% CI 45%-64%). Until now there is no well-established treatment for fatty liver disease.

Study setting: Randomized controlled trial

Study population:

Patients with type 2 DM plus Fatty Liver.

NAFLD diagnostic criteria:

* Fatty Liver Index (FLI) 60 or more plus Ultrasound features of fatty liver.

  - Inclusion criteria
  1. Age above 18. 2- HbA1C less than 10.

     Sample size: Based on the result reported by Armstrong et al, the proportion of patients on standard care who showed resolution of steatosis versus intervention group on liraglutide was 9% vs 39%, using power of 80%, precision of 5%, the minimal required sample size was 24 for each group and we increased it to 30 to compensate for drop-out. So, 120 subjects will be divided into 4 equal groups.

     Study Design: Interventional (Randomized Clinical Trial) Allocation: Randomized Intervention Model: Parallel Assignment Masking: No masking. Study duration: 12 months of follow up

     Data collection methods and tools

  <!-- -->

  1. Filling the pre-designed structured interview questionnaire from patients that includes:

     * Demographic traits: age, sex, marital status, education, occupation and residency.
     * Habits: smoking, physical exercise, dietary habits, drug use.
     * Social history, focusing on smoking status, occupation, presence of children at home and plans for future pregnancy (as appropriate).
     * Drug history
  2. Clinical data about:

     * Present/ past/ family history on thyroid diseases, and autoimmune disease.
     * Comorbidities: hypertension, coronary heart disease, chronic obstructive air way disease (COPD), obesity and others.
     * Medications used: dose, frequency and route of administration.
     * Hospitalization.
     * Body measures: weight, height, body mass index (BMI), waist circumference.
     * Vital signs: pulse, blood pressure, heart rate.
     * The compliance was ascertained through direct questioning at each clinic visits and by inspecting her pill bottles.
     * Patient satisfaction and quality of life will be measured at baseline and at the end of Intervention.
  3. Investigations

     * Lab: HCV Ab, HBsAg, HBcAb, ALT, AST, GGT, FBS, HBA1c, PPBS, Fasting insulin, CBC, Cholesterol, LDL, HDL, TGs, uric acid.
     * Calculation of the following score FLI, NAFLD-LFS, FIB-4, NFS.
     * Imaging: ultrasound/FIBROSCAN/ MRI.
     * Adverse effects of the drugs were systematically identified by careful health interview and clinical examinations. T-Bil, AST, ALT, and hematological values were measured for evaluation at every outpatient clinic visit.

     Follow-up

     All patients were followed up for twelve months:
* Dietary follow up.
* Liver enzymes (ALT, AST and GGT) at least every 3 months and more if clinically indicated
* Scores follow up: NFS and FIB-4 every 3 months.
* Fibroscan at end of 1-year follow up.
* MRI at end of 1-year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM with fatty liver disease.
* HbA1C less than 10.

Exclusion Criteria:

1. Alcohol intake.
2. BMI 40 or more.
3. CKD with e GFR less than 60.
4. chronic liver diseases (chronic viral hepatitis, autoimmune hepatitis, Wilson's disease, hemochromatosis, alfa-1 antitrypsin deficiency)
5. Atherosclerotic cardiovascular disease.
6. Celiac disease.
7. Clinically evident liver cirrhosis.
8. Patients who have ever had medullary thyroid carcinoma (MTC) or who have a family member who has ever had and patients who have multiple endocrine neoplasia syndrome type 2 (MEN 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in steatosis as measured using CAP score (fibroscan) and MRI | 12 months

SECONDARY OUTCOMES:
Change in liver enzymes | 12 months
Changes in fibrosis grade | 12 months
  as measured by transient elastography (Fibroscan)

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University., Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes